CLINICAL TRIAL: NCT03569657
Title: Activating Happiness in Cancer: A Positive Psychology Workshop for Patients, Survivors, and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Collaborators: Rocky Mountain Cancer Centers (Other)
Responsible Party: Principal Investigator, Trisha Raque-Bogdan, Assistant Professor, University of Denver
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1203830-2
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Caregivers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the group intervention, which is not part of routine medical care, to evaluate the group's effectiveness on participants' psychological well-being and their healthcare utilization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A positive psychology workshop (Other): The group intervention implements a manualized treatment protocol outlining the content of each of the four 90 minute sessions. The sessions will include topics such as mindfulness, self-compassion, gratitude and forgiveness, grief and growth, utilizing one's strengths, and resilience; with each session including homework exercises to be practiced between sessions. To assess the outcome measures, participants complete a baseline survey, a survey after the second session (2 weeks), a survey after the final session (4 weeks), and a follow-up survey 3 months after the workshop has ended (4 months).
  Interventions: Behavioral: A positive psychology workshop

INTERVENTIONS:
Behavioral: A positive psychology workshop — Group workshop

SUMMARY:
The number of worldwide cancer survivors is projected to be 21.3 million by 2030. To treat this growing population, group psychological interventions are increasingly utilized and require empirical support to evaluate their effectiveness. To address the need to assess positive group psychological interventions for cancer survivors and caregivers that incorporates diverse conceptualizations of adaption and examines both mental and physical health outcomes, this project is a study on a 4-week psychoeducation intervention group entitled "Activating happiness in cancer: A positive psychology workshop for patients, survivors, and caregivers." The project will evaluate the following hypotheses: (1) Participation in a positive psychology workshop will predict higher levels of well-being, mindfulness, gratitude, and vitality for cancer survivors and caregivers at the end of the group, and these changes will be maintained 3 months after the group has ended; and (2) Participation in a positive psychology intervention group will predict lower levels of depression, anxiety, pain, fatigue, loneliness, and healthcare utilization for cancer survivors and caregivers at the end of the group, and these changes will be maintained 3 months after the group has ended. Additionally, the project poses the following question: (1) What elements of positive psychological workshop do cancer survivors and caregivers perceive as most meaningful?

DETAILED DESCRIPTION:
The number of worldwide cancer survivors is projected to be 21.3 million by 2030. To treat this growing population, group psychological interventions are increasingly utilized and require empirical support to evaluate their effectiveness. Commonly reported psychosocial challenges that individuals face after a cancer diagnosis include depression, anxiety, pain, fatigue, and isolation. In contrast, some cancer survivors have reported increases in their sense of meaning, spirituality, and perceptions of personal growth after cancer. To address the range of responses to cancer, there is a need for strengths-based group interventions that optimize cancer survivors' psychosocial response to cancer, regardless of their distress level. It is critical for these approaches to account for normative periods of distress and despair for many cancer survivors, even as part of positive adaptation, and to honor "diversity in human response to cancer".

Cancer caregivers have reported similar clusters of symptoms as cancer survivors that often go untreated, in part due to the demands of caregiving responsibilities. Thus, cancer holds the potential to affect not only the patient, but also those closest in their social support network. Positive psychological interventions have demonstrated significant effects for increasing cancer survivors' self-esteem, optimism, self-efficacy, meaning making, and lowering levels of depression, anxiety, and fatigue. Yet no studies have examined the impact of positive psychological interventions on healthcare utilization, pain, loneliness, vitality, and self-compassion for cancer survivors, caregivers, and on the interactions between the well-being of cancer survivors and caregivers.

To address the need to assess positive group psychological interventions for cancer survivors and caregivers that incorporates diverse conceptualizations of adaption and examines both mental and physical health outcomes, this project is a study on a 4-week psychoeducation group intervention entitled "Activating happiness in cancer: A positive psychology workshop for patients, survivors, and caregivers." The project will evaluate the following hypotheses: (1) Participation in a positive psychology workshop will predict higher levels of well-being, mindfulness, gratitude, and vitality for cancer survivors and caregivers at the end of the group, and these changes will be maintained 3 months after the group has ended; and (2) Participation in a positive psychology workshop will predict lower levels of depression, anxiety, pain, fatigue, loneliness, and healthcare utilization for cancer survivors and caregivers at the end of the group, and these changes will be maintained 3 months after the group has ended. Additionally, the project poses the following question: (1) What elements of positive psychological workshop do cancer survivors and caregivers perceive as most meaningful? This intervention involves assigning participants to the group to evaluate its effectiveness on psychological and healthcare utilization outcomes. The group is not part of routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18
* either has received a cancer diagnosis OR
* is the caregiver of someone with a cancer diagnosis

Exclusion Criteria:

* Under the age 18
* Does not speak English
* Has not received a cancer diagnosis nor is the caregiver of someone with a cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Change in Depression | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Personal Health Questionnaire Depression Scale (Kroenke et al., 2009). "A total PHQ-8 score of 10 or greater in the clinical setting should prompt a careful interview for a number of reasons: to determine if the elevated score represents clinical depression, to consider confounding medical causes, to evaluate for affective disorders that may warrant either more conservative initial treatment than major depression (e.g., minor depression or bereavement) or earlier mental health referral (e.g., bipolar disorder or comorbid substance abuse), and to avoid premature labeling of a person as having depression."

SECONDARY OUTCOMES:
Change in Anxiety | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Generalized Anxiety and Depression (Spitzer, Kroenke, Williams, & Lowe, 2006). Scores are summed to get the total score, which can range from 0-21. Anxiety Severity Level:
  * Minimal: 0-4
  * Mild: 5-9
  * Moderate: 10-14
  * Severe: 15-21

OTHER OUTCOMES:
Change in Fatigue | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Multidimensional Fatigue Syndrome Inventory-Short Form (Stein, Jacobsen, Blanchard, & Thors, 2004). Score by summing individual subscales (General and Vigo subscales), ranging from 0 to 48. Higher scores indicate greater levels of fatigue.
  * General scale = sum of items 10, 12, 14, 17, 18, and 28
  * Vigor scale = sum of items 5, 7, 9, 22, 24, and 29
Change in Loneliness | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Three-Item Loneliness Scale (Hughes, Waite, Hawkley, & Cacioppo, 2008). Scores are summed to totaling all of the items, with a possible range from 0-9. Higher scores indicate higher levels of loneliness.
Change in Healthcare utilization | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Self-created questions asking how many times in the past week have you sought medical care that was not prescheduled. Items are not scored, and information is only being collected for background data.
Changes in Gratitude | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Gratitude Questionnaire-Six Item Form (McCullough, Emmons, & Tsang, 2002). To score, add up your scores for items 1, 2, 4, and 5. Add the reversed scores for items 3 and 6 to the total from Step 1. This is your total GQ-6 score. This number should be between 6 and 42. Higher scores indicate higher levels of gratitude.
Change in Mindfulness | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  State Mindfulness Scale (Tanay & Bernstein, 2013). Scores are totaled by summing all items, ranging from 21-105. Higher scores indicate higher levels of state mindfulness.
Change in Self-Compassion | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Self-Compassion Scale-Short Form (Neff, 2003). A total self-compassion score is computed by reversing the negative subscale items and then adding all subscale scores. Scores can range from 12-60, with higher scores indicating greater levels of self-compassion.
Change in Pain | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Brief Pain Inventory (Daut, Cleeland, & Flanery, 1983). Scores are summed to totaling all of the items, with a possible range from 0-50. Higher scores indicate more pain.
Change in Meaning in Life | Change from baseline to after 2nd session (2 weeks), baseline to after final session (4 weeks), baseline to after 3 months after final session (up to 16 weeks)
  Meaning in Life Questionnaire (Steger, Frazier, Oishi, & Kaler, 2006). Two subscales are totaled, one for the presence of life meaning (ranging from 0-35, higher levels indicate higher levels of life meaning) and one for the search for life meaning (ranging from 0-35, with higher levels indicating greater efforts directed at searching for life meaning).

CONTACTS AND LOCATIONS:
Locations (1):
- Rocky Mountain Cancer Centers, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No